CLINICAL TRIAL: NCT01190267
Title: A 26-week, Multi-center, Open-label, Flexible Dose, Long-term Safety Trial of Asenapine in Adolescent Subjects With Schizophrenia
Brief Title: Flexible Dose, Long-term Safety Study of Asenapine for the Treatment of Schizophrenia in Adolescents (P05897)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05897; 2009-018038-12 (EudraCT Number); MK-8274-021 (Other: Merck Research Laboratories)
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Results first posted 2014-08-06 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia, Paranoid; Schizophrenia, Disorganized; Schizophrenia, Undifferentiated
MeSH Terms: conditions — Schizophrenia, Paranoid; Schizophrenia, Disorganized; Schizophrenia; Disorders of Sex Development | interventions — asenapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Asenapine (Experimental): All enrolled participants receive open-label asenapine 2.5 mg twice daily (BID) on Day 1-3, which is increased to 5.0 mg BID on Day 4 (dose can be increased earlier at the investigator's discretion). Asenapine dosing is flexible for the remainder of the 26-week open-label drug administration period, and can be adjusted to either 2.5 mg or 5.0 mg BID at the investigator's discretion, based on tolerability and/or symptomatology.
  Interventions: Drug: asenapine

INTERVENTIONS:
Drug: asenapine — asenapine 2.5 mg or 5.0 mg sublingual tablets, administered BID
  Other Names: Saphris®, SCH 900274, Org 5222

SUMMARY:
This study is designed to evaluate whether asenapine, which is approved by the United States Food and Drug Administration (US FDA) for acute treatment of schizophrenia in adults, is generally safe and well tolerated in adolescents with schizophrenia. This is an extension of base study P05896 (NCT01190254), which means participants must have completed participation in the 8-week base study in order to qualify for this extension study P05897. Participants in this extension study will receive open-label asenapine for 26 weeks. Throughout the study, observations will be made on each participant at various times to assess the long-term safety, tolerability and efficacy of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must be between 12 and 17 years of age at the time of entry on this study, however, participants in the 8-week base study (P05896 [NCT01190254]) who reach 18 years of age while on P05896 may be enrolled in this extension study provided all other inclusion/exclusion criteria are met.
* Must have completed the 8-week efficacy and safety trial (P05896 [NCT01190254]) and, according to the investigator's judgment, would benefit from long-term treatment.
* Must have demonstrated an acceptable degree of compliance with trial medication, visits, and other requirements in the 8-week trial (P05896 [NCT01190254]), in the opinion of the investigator.

Exclusion Criteria:

* A female participant must not be pregnant and must not have the intention to become pregnant during the trial.
* A participant must not be at imminent risk of self-harm or harm to others.
* A participant must not currently be under involuntary inpatient commitment.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 204 (Actual)
Dates: Start 2010-09-28 (Actual); Primary Completion 2013-10-07 (Actual); Study Completion 2013-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Findling RL, Landbloom RP, Mackle M, Pallozzi W, Braat S, Hundt C, Wamboldt MZ, Mathews M. Safety and Efficacy from an 8 Week Double-Blind Trial and a 26 Week Open-Label Extension of Asenapine in Adolescents with Schizophrenia. J Child Adolesc Psychopharmacol. 2015 Jun;25(5):384-96. doi: 10.1089/cap.2015.0027. PMID 26091193

RESULTS

PARTICIPANT FLOW:
Groups:
- Asenapine - Participants Who Were ≤17 Years Old: In this extension study all participants received open-label asenapine 2.5 mg twice daily (BID) on Day 1-3, which was increased to 5.0 mg BID on Day 4 (dose could be increased earlier). Asenapine dosing was flexible for the remainder of the 26-week open-label drug administration period, and could be adjusted to either 2.5 mg or 5.0 mg BID. Participants in this reporting group were ≤17 years old at entry into the extension study.
- Asenapine - Participants Who Were 18 Years Old: In this extension study all participants received open-label asenapine 2.5 mg BID on Day 1-3, which was increased to 5.0 mg BID on Day 4 (dose could be increased earlier). Asenapine dosing was flexible for the remainder of the 26-week open-label drug administration period, and could be adjusted to either 2.5 mg or 5.0 mg BID. Participants in this reporting group were 18 years old at entry into the extension study.
Period: Overall Study
Arm/Group | Asenapine - Participants Who Were ≤17 Years Old | Asenapine - Participants Who Were 18 Years Old
Started | 196 | 8
Completed | 155 | 4
Not Completed | 41 | 4
Not completed — Adverse Event | 10 | 0
Not completed — Treatment Failure | 8 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 13 | 1
Not completed — Protocol Violation | 8 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of extension study medication
Groups:
- Asenapine - Participants Who Were ≤17 Years Old: In this extension study all participants received open-label asenapine 2.5 mg BID on Day 1-3, which was increased to 5.0 mg BID on Day 4 (dose could be increased earlier). Asenapine dosing was flexible for the remainder of the 26-week open-label drug administration period, and could be adjusted to either 2.5 mg or 5.0 mg BID. Participants in this reporting group were ≤17 years old at entry into the extension study.
- Total: Total of all reporting groups
Arm/Group | Asenapine - Participants Who Were ≤17 Years Old | Asenapine - Participants Who Were 18 Years Old | Total
Number analyzed (Participants) | 196 | 8 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (1.5) | 18 (0) | 15.4 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 4 | 78
  Male | 122 | 4 | 126

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Treatment-Emergent Adverse Event (AE) During Extension Study
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An AE was defined as a "treatment-emergent" AE if it was not present at the extension study baseline, or if it was present at the extension study baseline but worsened in severity compared to baseline during the extension study treatment period.
Time Frame: Up to 30 weeks
Population: All participants who received at least one dose of extension study medication
Measure: Number; unit: participants
Arm/Group | Asenapine - Participants Who Were ≤17 Years Old | Asenapine - Participants Who Were 18 Years Old
Number analyzed (Participants) | 196 | 8
participants | 114 | 3

2. Primary Outcome: Number of Participants Who Discontinued Study Drug During Extension Study Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Up to 26 weeks
Population: All participants who received at least one dose of extension study medication
Measure: Number; unit: participants
Arm/Group | Asenapine - Participants Who Were ≤17 Years Old | Asenapine - Participants Who Were 18 Years Old
Number analyzed (Participants) | 196 | 8
participants | 10 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 weeks
Description: The serious adverse events (SAEs) table includes all SAEs that occurred during this extension study. The Other AEs table includes only AEs in study that were "treatment-emergent" (i.e., not present at the extension study baseline, or present at the extension study baseline but worsened in severity compared to baseline during the extension study).
Arm/Group | Asenapine - Participants Who Were ≤17 Years Old | Asenapine - Participants Who Were 18 Years Old
Serious Adverse Events (participants affected / at risk) | 7/196 | 1/8
Other Adverse Events (participants affected / at risk) | 59/196 | 3/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine - Participants Who Were ≤17 Years Old (N=196) | Asenapine - Participants Who Were 18 Years Old (N=8)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 0 (0)
AGGRESSION (Psychiatric disorders) | 2 (2) | 0 (0)
AGITATION (Psychiatric disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 1 (1)
SCHIZOPHRENIA (Psychiatric disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine - Participants Who Were ≤17 Years Old (N=196) | Asenapine - Participants Who Were 18 Years Old (N=8)
VISION BLURRED (Eye disorders) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 5 (5) | 1 (1)
FEELING COLD (General disorders) | 0 (0) | 1 (1)
PAIN (General disorders) | 1 (1) | 1 (1)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 3 (4) | 1 (3)
INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
AKATHISIA (Nervous system disorders) | 4 (4) | 1 (1)
BRADYKINESIA (Nervous system disorders) | 0 (0) | 1 (1)
COGWHEEL RIGIDITY (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 13 (18) | 0 (0)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
RESTING TREMOR (Nervous system disorders) | 0 (0) | 1 (1)
SEDATION (Nervous system disorders) | 10 (11) | 1 (3)
SOMNOLENCE (Nervous system disorders) | 29 (36) | 0 (0)
TREMOR (Nervous system disorders) | 4 (4) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 3 (3) | 1 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ACNE (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is planned to first publish/present trial results together with the other sites, unless permission is obtained from Sponsor to publish separate results. Sponsor must be able to review all proposed results communications regarding study 45 days prior to submission for publication/presentation. If there is disagreement concerning appropriateness of the materials, Investigator and Sponsor must meet to make a good faith effort to discuss/resolve disagreement prior to submission for publication.